CLINICAL TRIAL: NCT03905044
Title: Clinical Characteristics of Three Pathological Types of Posterior Capsule Abnormality in Congenital Cataract Eyes
Brief Title: Clinical Characteristics in Congenital Cataract Eyes
Status: Completed | Type: Observational
Sponsor: yin ying zhao (Other)
Responsible Party: Sponsor-Investigator, yin ying zhao, Clinical professor, Wenzhou Medical University
Organization: Wenzhou Medical University (Other)
Other Study IDs: DXX-CC
Record Dates: First submitted 2019-04-03; First posted 2019-04-05 (Actual); Last update posted 2019-04-05 (Actual); Status verified 2019-04

CONDITIONS: Congenital Cataract
MeSH Terms: interventions — Vision, Ocular

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CC: eyes with congenital cataracts
  Interventions: Other: eyes with congenital cataracts

INTERVENTIONS:
Other: eyes with congenital cataracts — observation

SUMMARY:
This study involved children with congenial cataract eyes, who underwent cataract surgeries at the Eye Hospital of Wenzhou Medical University (Hangzhou, China). All medical records were reviewed for primary diagnosis. All surgeries were performed by one experienced surgeon (Z.Y.E) and videos were collected for reviews in details. the clinical data after the surgery were also recorded for further analysis.

ELIGIBILITY:
Inclusion Criteria:

* children with congenital cataracts who underwent cataract surgeries at the Eye Hospital of Wenzhou Medical University (Hangzhou, China)

Exclusion Criteria:

* ocular trauma

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: children with congenital cataracts
Sampling Method: Non-Probability Sample
Enrollment: 239 (Actual)
Dates: Start 2011-01-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
complication rate | 3 months
  the complication occurrent rate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ding X, Xiang L, Wang Q, Wang D, Chang P, Li Z, Zhao Y, Chu F, Ma C, Zhao YE. Clinical Characteristics and Surgical Safety in Congenital Cataract Eyes with Three Pathological Types of Posterior Capsule Abnormalities. J Ophthalmol. 2020 Mar 16;2020:6958051. doi: 10.1155/2020/6958051. eCollection 2020. PMID 32280529